CLINICAL TRIAL: NCT05360680
Title: A Phase 1, Open-Label, Dose Escalation and Expansion Study of CUE-102 Monotherapy in HLA-A*0201 Positive Patients With WT1 Positive Recurrent/Metastatic Cancers
Brief Title: A Phase 1 in Patients With HLA-A*0201+ and WT1+ Recurrent/Metastatic Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cue Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CUE-102-01
Record Dates: First submitted 2022-04-19; First posted 2022-05-04 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Gastric Cancer; Pancreatic Cancer; Ovarian Cancer
Keywords: Wilms' tumor 1; HLA A*0201
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Wilms Tumor

STUDY DESIGN:
Intervention Model Description: Phase 1 Dose Escalation and Expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CUE-102 (1mg/kg) Dose Escalation (Experimental): CUE-102 (1 mg/kg) Monotherapy IV infusion every 3 weeks for up to 2 years
  Interventions: Drug: CUE-102
- CUE-102 (2 mg/kg) Dose Escalation (Experimental): CUE-102 (2 mg/kg) Monotherapy IV infusion every 3 weeks for up to 2 years
  Interventions: Drug: CUE-102
- CUE-102 (4 mg/kg) Dose Escalation (Experimental): CUE-102 (4 mg/kg) Monotherapy IV infusion every 3 weeks for up to 2 years
  Interventions: Drug: CUE-102
- CUE-102 (8 mg/kg) Dose Escalation (Experimental): CUE-102 (8 mg/kg) Monotherapy IV infusion every 3 weeks for up to 2 years
  Interventions: Drug: CUE-102
- CUE-102 Dose Expansion at Determined RP2D (Experimental): Dose expansion of CUE-102 at determined RP2D Monotherapy IV infusion every 3 weeks for up to 2 years
  Interventions: Drug: CUE-102

INTERVENTIONS:
Drug: CUE-102 — CUE-102 is a novel fusion protein developed for the treatment of patients with WT1-positive malignancies.

SUMMARY:
This is a Phase 1, open-label, 2-part, multi-center study evaluating the safety, tolerability, PK, pharmacodynamics (PD), immunogenicity, and antitumor activity of CUE-102 intravenous (IV) monotherapy in HLA-A*0201 positive patients with WT1 positive recurrent/metastatic solid tumors who have failed conventional therapies.

DETAILED DESCRIPTION:
CUE-102 is a novel fusion protein developed for the treatment of patients with WT1-positive malignancies by selective engagement and expansion of tumor antigen-specific T cells that should allow for increased potential for anti-cancer efficacy and reduced toxicity relative to non-targeted forms of immunotherapy that result in systemic activation of the immune system.

The goal of Part A is to characterize the safety, tolerability, and biological effects of CUE-102.

The goal of Part B is to expand the safety and immune activity data at the RP2D identified in Part A, and to evaluate antitumor activity at this dose.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent and documentation of informed consent prior to initiation of any study-related tests or procedures that are not part of standard of care for the patient's disease.
2. Age ≥18 years old
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Life expectancy ≥12 weeks
5. Measurable disease as per RECIST 1.1 and documented by CT and/or MRI.
6. All tumors must have histologically or cytologically confirmed cancer diagnosis
7. Patients must have any of the following cancers to be eligible:

   A. Colorectal cancer
   1. Histologically or cytologically documented adenocarcinoma of colon or rectum at the time of initial presentation
   2. Metastatic or locally advanced/unresectable disease
   3. Documented disease progression after the last administration of standard therapies or intolerance to at least 2 prior systemic treatment regimens (CUE-102 will be 3rd line therapy or greater).

   B. Gastric cancer (including gastroesophageal junction)
   1. Histologically or cytologically documented gastric cancer at the time of initial presentation
   2. Metastatic or locally advanced/unresectable disease
   3. Documented disease progression after last administration of standard therapies or intolerance to standard therapies. (CUE-102 will be 2nd line therapy or greater).

   C. Pancreatic cancer
   1. Histologically or cytologically documented pancreatic adenocarcinoma at the time of initial presentation
   2. Patients with metastatic or locally advanced/unresectable disease.
   3. Prior systemic treatment must include either a fluoropyrimidine-based or gemcitabine-based regimen in either the (neo)adjuvant or relapsed setting. (CUE-102 will be 2nd line therapy or greater).

   D. Ovarian cancer
   1. Histologically or cytologically documented ovarian cancer at the time of initial presentation
   2. Metastatic or locally advanced/unresectable disease, with documented disease progression after last administration of standard therapies or intolerance to standard therapies.
   3. Prior systemic treatment must include a platinum-based regimen. (CUE-102 will be 2nd line therapy or greater).
   4. For patients determined to have platinum-sensitive disease, treatment with a second platinum-based combination regimen +/- bevacizumab should be considered prior to treatment with CUE-102 (CUE-102 will be 3rd line therapy or greater).
8. Patient must have HLA-A*0201 genotype as determined by genomic testing.
9. Patient must have histologically and/or cytologically proven tumor(s) that is WT1 positive.
10. Acceptable laboratory parameters.
11. Female patients of childbearing potential must agree to use acceptable contraceptive measures from the time of main study consent through 90 days after discontinuation of study drug administration.
12. Non-vasectomized male patients with partners of childbearing potential must use barrier contraception from the time of main study consent through 90 days after discontinuation of study drug.
13. Patients who have previously received an immune CPI (e.g., anti-programmed cell death ligand 1 (anti PD-L1), anti-programmed cell death 1 (anti-PD-1), anti-cytotoxic T lymphocyte-associated antigen 4 [CTLA-4]) prior to enrollment must have toxicities related to the CPI resolved to CTCAE ≤ Grade 1 or baseline (level prior to the CPI) to be eligible for enrollment. Patients who have experienced CPI-related endocrinopathies (e.g., diabetes, adrenal insufficiency) may participate if endocrinopathies are controlled (CTCAE ≤ Grade 1) with endocrinology support and appropriate repletion. Note: Patients who experienced previous hypothyroidism toxicity on a CPI are eligible to enter study regardless of CTCAE grade resolution as long as the patient is well controlled on thyroid replacement hormone.

Exclusion Criteria:

1. Female patients who are pregnant or plan to become pregnant during the course of the trial
2. Female patients who are breastfeeding
3. Patients with symptomatic central nervous system (CNS) metastases must have been treated, be asymptomatic, and not have any of the following at the time of enrollment:

   1. Need for concurrent treatment for the CNS disease (e.g., surgery, radiation, corticosteroids >10 mg prednisone/day or equivalent)
   2. Progression of CNS metastases on CT or MRI for at least 28 days after last day of prior therapy for the CNS metastases
   3. Concurrent leptomeningeal disease or cord compression.
4. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is permitted.
5. History of prior allogeneic bone marrow, stem-cell, or solid organ transplantation
6. Treatment with any systemic anti-neoplastic therapy, or investigational therapy within the 14 days (or 28 days, for antibody drugs), before the first dose of CUE-102.
7. Treatment with radiation therapy within 14 days before the first dose of CUE-102
8. Treatment with corticosteroids (> 10 mg per day prednisone or equivalent) or other immune suppressive drugs within 14 days before the first dose of CUE-102. Steroids for topical, ophthalmic, inhaled, or nasal administration are permitted. Physiological replacement with up to a maximum dose of 5 mg equivalence of prednisone per day is permitted.
9. History of clinically significant cardiovascular disease
10. Clinically significant pulmonary compromise (e.g., requirement for supplemental oxygen)
11. Clinically significant gastrointestinal (GI) disorders
12. Patients who experienced the following immune CPI-related AEs are ineligible even if the AE resolved to ≤ Grade 1 or baseline:

    1. ≥ Grade 3 ocular AE
    2. Changes in liver function tests that met the criteria for Hy's Law (> 3× ULN of either ALT/AST with concurrent > 2× ULN of total bilirubin (total and direct) and without alternate etiology)
    3. ≥ Grade 3 neurologic toxicity
    4. ≥ Grade 3 colitis
    5. ≥ Grade 3 renal toxicity
13. Evidence of active viral, bacterial, or systemic fungal infection requiring parenteral treatment within 7 days before the first dose of CUE-102.
14. No known history of infection or positive test for HIV, Hepatitis B or Hepatitis C, testing prior to enrollment is not required unless mandated by local authority
15. Second primary invasive malignancy that has not been in remission for > 2 years.
16. History of trauma or major surgery within 28 days before the first dose of CUE-102
17. Any serious underlying medical or psychiatric condition that would impair the ability of the patient to receive or tolerate the planned treatment at the investigational site
18. Known hypersensitivity to recombinant proteins, polysorbate 80 or any excipient contained in the drug formulation for CUE-102
19. Vaccination with any live virus vaccine within 28 days before the first dose of CUE-102. Inactivated annual influenza vaccination is allowed.
20. Dementia or altered mental status that would preclude understanding and rendering of informed consent
21. Active or history of significant alcohol or other substance abuse within 1 year before the first dose of CUE-102

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 21 Days
  Evaluate dose-limiting toxicities (DLTs) during the first cycle of treatment with CUE-102, and to establish a recommended Phase 2 dose (RP2D)
Maximum Tolerated Dose | 21 Days
  Evaluate maximum tolerated dose (MTD) to establish a recommended Phase 2 dose (RP2D)
Serum PK AUC for CUE-102 | Up to 2 years
  Area under the concentration-time curve (AUC) of CUE-102.
Serum PK Cmax for CUE-102 | Up to 2 years
  Maximum serum concentration (Cmax) of CUE-102.
Serum PK T1/2 for CUE-102 | Up to 2 years
  Terminal half-life (T1/2) of CUE-102.

SECONDARY OUTCOMES:
Safety and Tolerability of CUE-102 Assessed by NCI CTCAE v5.0 | Up to 2 years
  To evaluate safety and tolerability of CUE-102 using NCI CTCAE v5.0.
Antitumor Response Rate with Treatment of CUE-102 | Up to 2 years
  To evaluate antitumor response rate of CUE-102 by RECIST 1.1
Antitumor Duration of Response with Treatment of CUE-102 | Up to 2 years
  To evaluate antitumor duration of response of CUE-102 by RECIST 1.1
Antitumor Clinical Benefit Rate with Treatment of CUE-102 | Up to 2 years
  To evaluate antitumor clinical benefit rate of CUE-102 by RECIST 1.1
Progression-Free Survival with Treatment of CUE-102 | Up to 2 years
  To evaluate antitumor progression-free survival of CUE-102 by RECIST 1.1
Overall Survival with Treatment of CUE-102 | From First CUE-102 to Date of Death
  To evaluate overall survival after treatment with CUE-102
Immune Response Assessed by WW1 Tetramer-Positive T cell Lymphocytes | Up to 2 years
  To evaluate the potential for immune response after treatment with CUE-102 using assessment of number of WT1 tetramer-positive T cell lymphocytes.
Immune Response Assessed by CTL Markers of Activation | Up to 2 years
  To evaluate the potential for immune response after treatment with CUE-102 using assessment of cytotoxic T lymphocyte (CTL) markers of activation

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Levisetti, MD, Study Chair — Cue Biopharma
Locations (15):
- United States (15):
  - Mayo Clinic, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford Advanced Medicine Cancer Center, Palo Alto, California
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Carol G. Simon Cancer Center - Morristown Medical Center, Morristown, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Cleveland Medical Center (University Hospitals), Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - Carbone Cancer Center, Madison, Wisconsin